CLINICAL TRIAL: NCT06388681
Title: The Effect of Stress Ball Use on Immobilization Comfort, Pain Level and Vital Signs in Patients Undergoing Coronary Angiography
Brief Title: Stress Ball Use in Patients Undergoing Coronary Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Sumeyye Akcoban, Principal Investigator, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HMKU-KMY-SA-02
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Pain
Keywords: Pain; Vital Signs; Patient Comfort; Angiography
MeSH Terms: conditions — Pain | interventions — Vital Signs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Intervention Group Patients in the intervention group will be allowed to use a stress ball. The comfort level, vital signs and pain intensity of the patients in the intervention group will be evaluated with the Immolization comfort scale 2 hours before Sheath extraction. Pain intensity and vital signs will be evaluated 2 hours after sheath extraction, and comfort level, vital signs and pain intensity will be evaluated with Immolization comfort scale 4 hours after sheath extraction.
  Stress Ball Use Practice for the Intervention Group The researchers will explain and demonstrate to the intervention group how to use the stress ball. Then, the patient will be asked to use the ball and it will be confirmed whether he/she uses it correctly. After angiography, it will be stated that the patients in the intervention group should count to 5 and squeeze it once for 10 minutes every hour and rotate with the right and left hand until they are mobilized.
  Interventions: Device: The Effect of Stress Ball Use on Immobilization Comfort, Pain Level and Vital Signs in Patients Undergoing Coronary Angiography
- Control Group (No Intervention): Control Group Patients in the control group will not undergo any intervention. Comfort level, vital signs and pain will be evaluated with Immolization comfort scale 2 hours before Sheath extraction. Pain and vital signs will be evaluated 2 hours after Sheath extraction and comfort level, vital signs and pain will be evaluated with Immolization comfort scale 4 hours after Sheath extraction.

INTERVENTIONS:
Device: The Effect of Stress Ball Use on Immobilization Comfort, Pain Level and Vital Signs in Patients Undergoing Coronary Angiography — The researchers will explain and demonstrate to the intervention group how to use the stress ball. Then, the patient will be asked to use the ball and it will be confirmed whether he/she uses it correctly. After angiography, it will be stated that the patients in the intervention group should count to 5 and squeeze it once for 10 minutes every hour and rotate with the right hand and left hand until they are mobilized.
  Arms: Experimental

SUMMARY:
One of the nonpharmacologic interventions included in the NIC-Nursing Interventions Classification is the use of stress balls. Stress balls are one of the cognitive distraction methods used especially in reducing pain and increasing the comfort level of patients. On the other hand, there are studies showing that stress balls have a positive effect not only on pain but also on vital signs, anxiety and comfort level of the patient.

DETAILED DESCRIPTION:
The study will be conducted in the cardiology clinics of a state hospital between April 2024 and June 2024. The study was planned as a randomized experimental study to examine the effect of stress ball use on immobilization comfort, pain level and vital signs in patients undergoing coronary angiography. The population of the study consisted of patients admitted to the cardiology clinic of a state hospital. G*Power 3.1.9.7 program was used for sample size calculation. Cohen's standardized effect size was used since no study with similar sample characteristics and criteria was found. Friedman's F Test was used to evaluate whether the effect on immobilization comfort, pain level and vital signs differed between the intervention and control groups of patients undergoing angiography through the femoral artery. Accordingly, the sample size was determined as (n=66), intervention group (n=33), control group (n=33) with a low effect size (0.2) in line with the relevant tests and a pyori calculation with α error=0.05, (1-β error) =0.95. A total of 72 patients, 36 in each group, were planned to be included in the study with a 10% patient loss. The patient information form prepared by the investigators will be filled in before transfer to the angiography procedure room for the patients who were determined as intervention (n=36) and control group (n=36). Data will be evaluated in 3 stages: 2 hours before sheath extraction, 2 hours after sheath extraction and 4 hours after sheath extraction. The researchers will explain and demonstrate to the intervention group how to use the stress ball. Then, the patient will be asked to use the ball and it will be confirmed whether they use it correctly. After angiography, it will be stated that the patients in the intervention group should count to 5 and squeeze it once for 10 minutes every hour and rotate with the right and left hand until they are mobilized. The stress ball used will be of medium hardness and made of high quality silicone. Stress balls will be provided by the researchers and given to the patients. Patients in the control group will not undergo any intervention. Comfort level, vital signs and pain will be evaluated with Immolization comfort scale 2 hours before Sheath extraction. Pain and vital signs will be evaluated 2 hours after Sheath extraction and comfort level, vital signs and pain will be evaluated with Immolization comfort scale 4 hours after Sheath extraction.

ELIGIBILITY:
Inclusion Criteria:

* Who are over 18 years old,
* Having no barriers to written and verbal communication in Turkish,
* Patients without chronic dermatological and/or vascular disease
* Patients undergoing angiography via the femoral artery will be included in the trial

Exclusion Criteria:

* Patients who cannot communicate verbally
* Patients with a psychiatric diagnosis
* Patients who drop out of the study at any stage of the study
* Patients who underwent angiography using an artery other than the femoral artery will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Immobilization Comfort Scale | Comfort assessment with Immobilization Comfort Scale will be performed 2 hours before, 2 hours and 4 hours after sheath extraction.
  The Turkish validity and reliability study of the scale developed by Hogan-Miller in 1995 was conducted. The scale consists of 20 items. Each statement in the scale has a Likert-type scoring ranging from 1-6 from "strongly disagree" to "strongly agree". Items 2, 3, 4, 7, 8, 10, 13, 14 and 18 in the scale are negative statements. The total scores obtained from the scale vary between 20 and 120, with a high score indicating good comfort. Cronbach's alpha value of the scale was found to be 0.82.
Visual Benchmarking Scale | Pain assessment will be performed with Visual Comparison Scale 2 hours before, 2 hours and 4 hours after sheath extraction.
  The scale allows patients to measure their own pain level by marking their pain level on a 10 cm ruler at intervals ranging from "no pain" to "most severe pain". The scale has been reported to be more sensitive and reliable than other unidimensional scales in measuring pain level. A study was conducted to standardize this scale and it was found that the vertical use of the scale was better understood by patients. In this model, the patient is told that "the scale has two endpoints and he/she is free to mark any point between these points that corresponds to his/her pain level". The interval between the "pain-free" point and the point marked by the patient is recorded in centimeters using a ruler.

SECONDARY OUTCOMES:
Nurse Observation Form | 2 hours before the sheath extraction, 2 hours and 4 hours after the sheath extraction; vital signs will be evaluated with the vital signs recorded on the Nurse Observation Form.
  Vital signs (Blood Pressure, Pulse, Temperature, Respiration and Partial Oxygen Pressure) will be taken from the nurse observation form recorded every hour.

CONTACTS AND LOCATIONS:
Overall Officials: SÜMEYYE AKÇOBAN, Principal Investigator — Mustafa Kemal University
Locations (1):
- Hatay Mustafa Kemal University, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Genc H, Korkmaz M, Akkurt A. The Effect of Virtual Reality Glasses and Stress Balls on Pain and Vital Findings During Transrectal Prostate Biopsy: A Randomized Controlled Trial. J Perianesth Nurs. 2022 Jun;37(3):344-350. doi: 10.1016/j.jopan.2021.09.006. Epub 2022 Apr 7. PMID 35397973
- [Background] Rejeh N, Tadrisi SD, Yazdani S, Saatchi K, Vaismoradi M. The Effect of Hand Reflexology Massage on Pain and Fatigue in Patients after Coronary Angiography: A Randomized Controlled Clinical Trial. Nurs Res Pract. 2020 Aug 29;2020:8386167. doi: 10.1155/2020/8386167. eCollection 2020. PMID 32908698
- [Derived] Akcoban S, Tosun B, Yuksel H. The Effect of Stress Ball Use on Immobilization Comfort, Pain Level, and Vital Signs in Patients After Coronary Angiography. J Cardiovasc Nurs. 2026 Jan-Feb 01;41(1):E25-E32. doi: 10.1097/JCN.0000000000001202. Epub 2025 Apr 9. PMID 40198758